CLINICAL TRIAL: NCT01048879
Title: Pharmacokinetics of Tamiflu® (Oseltamivir) in Patients Receiving CVVHD and/or ECMO
Brief Title: Pharmacokinetics of Tamiflu® (Oseltamivir) in Patients Receiving Extracorporeal Membrane Oxygenation (ECMO)and or Continuous Venovenous Hemodialysis (CVVHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Bruce A. Mueller, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00033929
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Critically Ill Renal Failure Requiring CVVHD and Oseltamivir; Critically Ill Requiring ECMO and Oseltamivir
Keywords: oseltamivir; influenza; continuous renal replacement therapy; extracorporeal membrane oxygenation; pharmacokinetics
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ECMO alone (Other): Patients receiving oseltamivir and Extracorporeal Membrane Oxygenation (ECMO) therapy (patients were already receiving oseltamivir and ECMO due to an illness)- Procedure/Surgery: pharmacokinetic blood sampling
  Interventions: Procedure: pharmacokinetic blood sampling
- CVVHD Alone (Other): Patients receiving Continuous Venovenous Hemodialysis(CVVHD) and oseltamivir (Patients were already receiving oseltamivir and CVVHD as a result of an illness).
  Procedure/Surgery: pharmacokinetic blood and dialysate sampling
  Interventions: Procedure: pharmacokinetic blood and dialysate sampling
- CVVHD + ECMO (Other): Patient receiving oseltamivir and ECMO and CVVHD (patients were already receiving oseltamivir, ECMO, and CVVHD as part of an illness).
  Procedure/Surgery: pharmacokinetic blood and dialysate sampling
  Interventions: Procedure: pharmacokinetic blood and dialysate sampling

INTERVENTIONS:
Procedure: pharmacokinetic blood sampling — blood samples collected to assess oseltamivir concentrations
  Other Names: Tamiflu
  Arms: ECMO alone
Procedure: pharmacokinetic blood and dialysate sampling — blood and dialysate samples collected and assayed for oseltamivir concentrations
  Other Names: Tamiflu
  Arms: CVVHD + ECMO; CVVHD Alone

SUMMARY:
Critically ill patients with flu may receive a drug called oseltamivir. They may also receive medical therapies to support their lung function (extracorporeal membrane oxygenation; ECMO) and kidney function (continuous venovenous hemodialysis; CVVHD). CVVHD and ECMO may remove some oseltamivir from the bloodstream. The purpose of this study is to determine how much oseltamivir gets removed by CVVHD or ECMO in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* receiving Continuous Venovenous Hemodialysis (CVVHD) or Extracorporeal Membrane Oxygenation (ECMO)
* require oseltamivir treatment
* informed consent granted

Exclusion Criteria:

* pregnant
* unable to complete 12 hours of CVVHD or ECMO
* <6 kg body weight
* allergy to oseltamivir

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Mueller, Pharm.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Eyler RF, Heung M, Pleva M, Sowinski KM, Park PK, Napolitano LM, Mueller BA. Pharmacokinetics of oseltamivir and oseltamivir carboxylate in critically ill patients receiving continuous venovenous hemodialysis and/or extracorporeal membrane oxygenation. Pharmacotherapy. 2012 Dec;32(12):1061-9. doi: 10.1002/phar.1151. PMID 23208833

RESULTS

PARTICIPANT FLOW:
Groups:
- ECMO Alone: Patients receiving oseltamivir and Extracorporeal Membrane Oxygenation (ECMO) therapy
- CVVHD Alone: Patients receiving Continuous Venovenous Hemodialysis(CVVHD) and oseltamivir
- CVVHD + ECMO: Patient receiving oseltamivir and ECMO and CVVHD
Period: Overall Study
Arm/Group | ECMO Alone | CVVHD Alone | CVVHD + ECMO
Started | 1 | 9 | 5
Completed | 1 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ECMO Alone | CVVHD Alone | CVVHD + ECMO | Total
Number analyzed (Participants) | 1 | 9 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 1 | 8 | 4 | 13
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (0) | 33.0 (10.2) | 32.2 (16.1) | 33.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 4
  Male | 1 | 6 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 1 | 9 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Continuous Venovenous Hemodialysis (CVVHD)Oseltamivir Carboxylate Transmembrane Clearance
Description: Oseltamivir Carboxylate Transmembrane Clearance by Continuous Venovenous Hemodialysis (Reported in mL/min).
Time Frame: 12 hours
Population: One patient in the CVVHD Alone group was excluded from the analysis because not enough data points were available for pharmacokinetic modeling.
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- CVVHD + ECMO: Patients receiving oseltamivir and ECMO and CVVHD
- ECMO Alone: Patients receiving ECMO only
Arm/Group | CVVHD Alone | CVVHD + ECMO | ECMO Alone
Number analyzed (Participants) | 8 | 5 | 0
mL/min | 52.2 (8.0) | 43.3 (6.7) |

2. Primary Outcome: Oseltamivir Carboxylate Removal by ECMO
Description: Mean percent change in oseltamivir carboxylate concentration pre- and post-oxygenator.
Time Frame: 12 hours
Population: All of the patients that received ECMO were included. Patients receiving CVVHD Alone did not receive ECMO and were not included.
Measure: Mean (Standard Deviation); unit: percent change in concentration
Arm/Group | CVVHD Alone | CVVHD + ECMO | ECMO Alone
Number analyzed (Participants) | 0 | 5 | 1
percent change in concentration |  | -0.008 (0.101) | -0.033 (0.082)

ADVERSE EVENTS:
Arm/Group | ECMO Alone | CVVHD Alone | CVVHD + ECMO
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No